CLINICAL TRIAL: NCT05335928
Title: AbatacepT foR ImmUne Checkpoint Inhibitor Associated Myocarditis (ATRIUM): A Phase 3, Investigator-Initiated, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Abatacept in ICI Myocarditis
Brief Title: Abatacept in Immune Checkpoint Inhibitor Myocarditis
Acronym: ATRIUM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Tomas G. Neilan, MD, Director, Cardio-Oncology Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P003690
Record Dates: First submitted 2022-04-05; First posted 2022-04-20 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Myocarditis Acute; Cancer
Keywords: Immune checkpoint Inhibitor; Myocarditis; Abatacept; Immune therapy; Immune related adverse events
MeSH Terms: conditions — Neoplasms; Myocarditis | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abatacept plus standard of care (Experimental): Abatacept (10 mg/kg) will be administered IV after randomization, again at 24 hours after first study drug treatment, at 14 days after first study drug treatment and an optional 4th dose at 28 days.
  Interventions: Drug: Abatacept plus
- Placebo plus standard of care (Placebo Comparator): Placebo will be administered at the same intervals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept plus — Up to 4 study drug infusions at 10 mg/kg, IV
  Drug: Standard of care Local standard of care per written policies or guidelines Other Name: SoC
  Other Names: Orencia
  Arms: Abatacept plus standard of care
Drug: Placebo — Drug: Standard of care Local standard of care per written policies or guidelines Other Name: SoC
  Arms: Placebo plus standard of care

SUMMARY:
The primary aim is to test whether abatacept, as compared to placebo, is associated with a reduction in major adverse cardiac events (MACE) among participants hospitalized with myocarditis secondary to an immune checkpoint inhibitor (ICI). The primary outcome, MACE, is a composite of first occurrence of cardiovascular death, non-fatal sudden cardiac arrest, cardiogenic shock, significant ventricular arrythmias, significant bradyarrythmias, or incident heart failure.

DETAILED DESCRIPTION:
This investigator-initiated randomized trial is being conducted to test whether abatacept, as compared to placebo, is associated with a reduction in MACE among participants who develop myocarditis after treatment with an ICI. Immune checkpoint inhibitors leverage the immune system to treat a wide variety of cancers. Myocarditis is an uncommon immune related adverse event (irAE) secondary to treatment with an ICI. The guideline recommended treatment for ICI myocarditis is cessation of the ICI and administration of corticosteroids. However, despite administration of corticosteroids, the rate of MACE with ICI myocarditis is high. Data from multiple independent international cohorts have shown that the rate of MACE with ICI myocarditis despite administration of corticosteroids ranges from 25-50%.For comparison, the rate of MACE with myocarditis unrelated to an ICI is <5%.

Abatacept is a selective co-stimulation modulator that inhibits T cell (T lymphocyte) activation by binding to CD80 and CD86, thereby blocking its interaction with CD28. This interaction provides a costimulatory signal necessary for full activation of T lymphocytes. In animal studies of ICI myocarditis, the administration of abatacept led to a reduction in cardiac immune activation and an increase in survival. In retrospective unpublished clinical data, the administration of abatacept to participants with ICI myocarditis on corticosteroids was associated with a reduction in risk of MACE. There are no prospective studies testing whether abatacept is effective among participants with ICI myocarditis. Therefore, the primary aim of this trial is to test in a randomized double-blind placebo-controlled study whether abatacept, administered concurrently with corticosteroids, is associated with a reduction in MACE among participants with recently diagnosed ICI myocarditis

ELIGIBILITY:
Inclusion Criteria:

1. Must have provided informed consent in a manner approved by the Investigator's Institutional Review Board (IRB) prior to any study-related procedure being performed. If a participant is unable to provide informed consent due to his/her medical condition, the participant's legally authorized representative may consent on behalf of the study participant, as permitted by local law and institutional Standard Operating Procedures;
2. Aged greater than or equal to 18 years at the time of informed consent;
3. Recent use of an FDA-approved immune checkpoint inhibitor (ICI, defined as administered an immune checkpoint inhibitor ≤ 6 months of myocarditis diagnosis), alone or in combination with other cancer therapies (i.e. chemotherapy, radiation therapy or targeted therapy). The FDA-approved ICI could be given as part of a clinical trial but not in combination with a new investigational agent which may cause myocarditis;
4. A diagnosis of myocarditis.
5. Hospitalized at the time of randomization;
6. On 1000 mg of solumedrol per day for myocarditis or with an intent to initiate 1000 mg of solumedrol per day for myocarditis within 24 hours of first administration of study drug;
7. Serum evidence of ongoing myocardial injury: Serum evidence of ongoing myocardial injury will be defined as an institutional troponin (either conventional or high-sensitivity troponin I or T, using the standard institutional assay) with a value that is ≥5 times the upper limit of the reference standard normal for that institution. The troponin assay may be adjusted based on sex depending on institutional standards. This value of troponin of ≥5 times above the institutional upper limits of normal value must be noted within 10 days prior to potential randomization. The 10-day period can be in the outpatient or inpatient setting. For example, a participant with a troponin value that on one occasion was ≥5 times the upper limits of institutional normal in the 10-day window prior to potential randomization (whether in the inpatient or outpatient setting), but later decreases below that threshold, typically due to starting corticosteroids, would still be considered eligible;
8. The following laboratory parameters, not older than 48 hours at the time of randomization, and measured as part of usual care:

   * Total white blood cell (WBC) count >2,500/μl
   * Absolute neutrophil count (ANC) >1,500/μL
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) <20 times the upper limit of the institutional normal ranges;
9. Women of childbearing potential (i.e., not postmenopausal, or surgically sterilized) must have a negative highly sensitive urine or serum pregnancy test prior to randomization. Participating women of childbearing potential must be willing to consistently use effective methods of contraception from screening until at least 90 days after administration of the last dose of study drug. Participating men must also be willing to consistently use effective methods of contraception from screening until at least 90 days after administration of the last dose of study drug; and
10. Must be willing and able to abide by all study requirements and restrictions.

Exclusion Criteria:

1. Must not have experienced any of the following (as defined in the section on the primary endpoint) in the 30-day period prior to randomization:

   * A sudden cardiac arrest
   * Cardiogenic shock as defined. A significant bradyarrhythmia (Mobitz type II second degree atrioventricular block or third degree (complete) atrio-ventricular (AV) block, for which an intervention with a temporary or permanent pacemaker is completed or recommended).
   * A significant tachyarrhythmia (ventricular fibrillation of any duration or sustained ventricular tachycardia (>30 seconds, >120 beats per minute); or a ventricular tachyarrhythmia requiring intervention.
2. Recent (≤2 month) exposure to abatacept or belatacept.
3. Concurrent or recent (≤2 month) use of the following non-corticosteroid immunosuppressive therapies prior to randomization: mycophenolate, JAK STAT inhibitors (including but not limited to upadacitinib, tofacitinib, baricitinib, and filgotinib), tacrolimus, anti-thymocyte globulin, alemtuzumab, infliximab, and plasma exchange. The use of intravenous immunoglobulin is permitted prior to randomization and during study treatment.
4. Currently enrolled in another interventional study utilizing systemic agents for the management of ICI-related toxicities.
5. Female who is pregnant, breastfeeding, or is considering becoming pregnant during the study or for approximately 90 days after the last dose of study drug.
6. Male who is considering fathering a child or donating sperm during the study or for approximately 30 days after the last dose of study drug.
7. Any active, chronic, or recurrent viral infection that, based on the investigator's clinical assessment, makes the participant an unsuitable candidate for the study. These may include hepatitis B virus (HBV) or hepatitis C virus (HCV), recurrent or disseminated (even a single episode) herpes zoster, and disseminated (even a single episode) herpes simplex. Active HBV and HCV are defined as: HBV: hepatitis B surface antigen (HBs Ag) positive (+) or detected sensitivity on the HBV deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) qualitative test for Hepatitis B core antibody (HBc Ab) positive (+) participants; HCV: HCV ribonucleic acid (RNA) detectable in any participant with anti-HCV antibody (HCV Ab). Patients with active Covid-19 infection will be excluded. This is defined as the period of ongoing symptoms in the setting of a positive Covid-19 test, or until 10 days after symptom onset and after resolution of fever for at least 24 hours, without the use of fever-reducing medications.
8. Known active tuberculosis (TB), history of incompletely treated TB, suspected or known extrapulmonary TB, suspected or known systemic bacterial or fungal infections;
9. Receipt of any live vaccine within four weeks prior to the first dose of study drug, or expected need of live vaccination during study participation including at least 90 days after the last dose of IV study drug.
10. Any medical condition that could interfere with, or for which the treatment might interfere with, the conduct of the study or interpretation of the study results, or that would, in the opinion of the Investigator, increase the risk of the participant by participating in the study.
11. Any factors that, in the Investigator's opinion, are likely to interfere with study procedures, such as history of noncompliance with scheduled appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2022-07-02 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-04-20 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 6 months
  The rates of a composite of cardiovascular death, non-fatal sudden cardiac arrest, cardiogenic shock, significant ventricular arrhythmias, significant bradyarrhythmias, or incident heart failure.

SECONDARY OUTCOMES:
The individual components of the primary endpoint. | 6 months
  The rates of the following between groups: cardiovascular death, non-fatal sudden cardiac arrest, cardiogenic shock, significant ventricular arrhythmias, significant bradyarrhythmias, or incident heart failure
Myocarditis illness severity using a 7-point ordinal severity scale containing each of the individual endpoints in a hierarchical ranking order. | 6 months
  The worst score on a 7-point ordinal myocarditis severity scale during the 6 month period from first study treatment. The 7-point ordinal myocarditis severity scale is as follows with more severe outcomes ranked with a higher number:
  1. - No component of the primary endpoint;
  2. - Incident heart failure;
  3. - Significant bradyarrhythmia;
  4. - Significant ventricular tachyarrhythmias;
  5. - Cardiogenic shock;
  6. - Sudden cardiac arrest;
  7. - Cardiovascular death;
The increase in serum troponin levels | 6 months
  The proportion of participants in each group with a >50% increase in serum troponin value at any time during the incident hospitalization and following administration of study drug.
The combination of the rates of the primary outcome plus the proportion of patients with a troponin increase. | 6 months
  The rates of a composite of cardiovascular death, non-fatal sudden cardiac arrest, cardiogenic shock, significant ventricular arrhythmias, significant bradyarrhythmias, or incident heart failure plus the proportion of participants in each group with a >50% increase in serum troponin value at any time during the incident hospitalization and following administration of study drug.
Clinical status at 90 days after first infusion of study drug | 6 months
  Clinical status at visit 6 (day 90) on an ordinal scale with highest being the worst:
  1. - Alive and off corticosteroids for myocarditis;
  2. - Alive and on corticosteroids (provide dose) for myocarditis;
  3. - Alive and on cellcept (provide dose) for myocarditis;
  4. - Alive and on both corticosteroids (provide dose) and cellcept (provide dose) for myocarditis
  5. - Dead (cancer, cardiovascular or other).
Clinical status at 6 months after first infusion of study drug | 6 months
  Clinical status at visit 7 (6 months) with the highest being the worst:
  1. - Alive and off corticosteroids for myocarditis;
  2. - Alive and on corticosteroids (provide dose) for myocarditis;
  3. - Alive and on cellcept (provide dose) for myocarditis;
  4. - Alive and on both corticosteroids (provide dose) and cellcept (provide dose) for myocarditis
  5. - Dead (cancer, cardiovascular or other).
Fatal and non-fatal DVT and PE | 6 months
  The proportion of patients in each group with a fatal and non-fatal DVT and PE will be compared.
Other immune-related adverse events between the two groups | 6 months
  Rates of other immune-related adverse events between the two groups will be compared.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (29):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - MedStar Health Research Institute, Georgetown University, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Franciscan Health, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Maine Health, Portland, Maine
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Lehigh Valley Health Network, Bethlehem, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institution, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of West Virginia, Morgantown, West Virginia
  - Aurora St Luke's Medical Center, Milwaukee, Wisconsin
- Canada (2):
  - University of British Colombia, Vancouver, British Colombia
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Heymans S, Van Linthout S, Kraus SM, Cooper LT, Ntusi NAB. Clinical Characteristics and Mechanisms of Acute Myocarditis. Circ Res. 2024 Jul 5;135(2):397-411. doi: 10.1161/CIRCRESAHA.124.324674. Epub 2024 Jul 4. PMID 38963866